CLINICAL TRIAL: NCT04045730
Title: A Single Arm Phase 2 Study of Gemcitabine Plus Nab-Paclitaxel in Combination With Pegvorhyaluronidase Alfa (PVHA; PEGPH20) and Pembrolizumab as Front-line Treatment for Metastatic Pancreatic Adenocarcinoma.
Brief Title: The Study of Gemcitabine Plus Nab-Paclitaxel in Combination With Pegvorhyaluronidase Alfa (PVHA; PEGPH20) and Pembrolizumab as Front-line Treatment for Metastatic Pancreatic Adenocarcinoma.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Halozyme isn't allowing this trial to move forward until their current clinical trial results are released.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000024450
Record Dates: First submitted 2019-07-02; First posted 2019-08-05 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Pancreas Adenocarcinoma
MeSH Terms: interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is an open-label single arm
Masking Description: This is an open-label single arm
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with metastatic pancreatic ductal adenocarcinoma (Experimental): Patients must have histologically or cytologically confirmed pancreatic ductal adenocarcinoma, and all patients must have at least 15 unstained slides of formalin fixed paraffin embedded (FFPE) tumor tissue available or a pre-treatment core needle biopsy will be required as outlined in section 7.1.2.7. All patients will receive treatment with gemcitabine, nab-paclitaxel, PVHA, and pembrolizumab in 4-week cycles.
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Gemcitabine — All patients will receive treatment with gemcitabine, nab-paclitaxel, PVHA, and pembrolizumab.
  Other Names: nab-paclitaxel; PVHA; pembrolizumab

SUMMARY:
This is an open-label single arm phase 2 study for patients with metastatic pancreatic ductal adenocarcinoma who have not received any prior systemic therapies.

DETAILED DESCRIPTION:
To determine the efficacy of gemcitabine plus nab-paclitaxel in combination with PVHA and pembrolizumab as measured by progression free survival (PFS).

Hypothesis: The combination of gemcitabine, nab-paclitaxel, PVHA and pembrolizumab will improve PFS compared to the historical control for chemotherapy.

3.2 Secondary Objectives & Hypotheses

1. Objective: To estimate median overall survival (OS)
2. Objective: To determine the overall response rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
3. Objective: To determine the toxicity and tolerability of gemcitabine plus nab-paclitaxel with PVHA and pembrolizumab.

Hypothesis: The combination of gemcitabine, nab-paclitaxel, PVHA, and pembrolizumab will be safe and improve OS and ORR compared to the historical control for chemotherapy.

3.3 Exploratory Objective

1. Objective: To evaluate pre-treatment and on-treatment PD-L1 and hyaluronan (HA) status and correlate with PFS, ORR, and OS.
2. Objective: To measure the stromal alterations and stromal degradation of hyaluronan and correlate with clinical benefit.
3. Objective: To quantify the pre-treatment and on-treatment change in immune effector cells and correlate with clinical benefit.
4. Objective: To cryopreserve additional tumor tissue for future analysis, including but not limited to DNA and RNA sequencing.
5. Objective: To create organoid cultures from core biopsy specimens for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Male/female participants who are at least 18 years of age on the day of signing informed consent with an untreated metastatic histologically confirmed diagnosis of stage IV pancreatic ductal adenocarcinoma will be enrolled in this study.
* Male participants:

A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.

* Female participants:

A female participant is eligible to participate if she is not pregnant not breastfeeding, and at least one of the following conditions applies: Not a woman of childbearing potential (WOCBP) as defined in Appendix 3

A WOCBP who agrees to follow the contraceptive guidance in during the treatment period and for at least 120 days after the last dose of study treatment.

* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial. Patients or their legally authorized representative must be informed of the investigational nature of this study.
* Measurable disease on computed tomography (CT) scan and/or MRI per RECIST 1.1 criteria. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Willing to undergo a pre-treatment core or excisional biopsy of a tumor lesion not previously irradiated, except for patients with 15 FFPE unstained slides of tumor tissue where a pre-treatment biopsy is optional. If 15 FFPE unstained slides are unavailable a pre-treatment biopsy is only mandatory if it can be obtained via a non-significant risk procedure. Significant risk procedures include (but are not limited to) biopsies of the brain, lung / mediastinum, pancreas, or endoscopic procedures extending beyond the esophagus, stomach, or bowel. Any biopsy via significant risk procedure is optional. For patients who pursue an optional biopsy when a non-significant risk biopsy is possible the optional biopsy will serve as the pre-treatment tissue sample. Biopsy requirements are further outlined in section 7.1.2.7.
* Willing to undergo an on-treatment core or excisional tumor biopsy at week 8 (for the first 20 evaluable patients). Biopsy risk requirements for on-treatment biopsies are the same as the pre-treatment biopsy and outlined above and in section 7.1.2.7.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to day 1 of treatment. .
* Has a life expectancy of ≥ 20 weeks.
* Has adequate organ function as defined in the following table (Table 1). Specimens must be collected within 10 days prior to the start of study treatment.

Exclusion Criteria:

* A WOCBP who has a positive urine pregnancy test within 72 hours prior to the first dose of study treatment (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Has received any prior systemic anti-cancer therapy including investigational agents for their metastatic pancreatic ductal adenocarcinoma prior to the first dose of study treatment. This includes any patients that have progressed ≤ 6 months of adjuvant therapy.

Note: Participants must have recovered from all Adverse Events (AE) due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible.

Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.

* Has received any prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), OX40, CD137).
* Has received prior radiotherapy for metastatic pancreatic ductal adenocarcinoma prior to the first dose of study treatment.
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Has known history of Central Nervous System (CNS) metastases and/or carcinomatous meningitis, regardless of whether or not they have been treated.
* Has severe hypersensitivity (≥Grade 3) to gemcitabine, nab-paclitaxel, PVHA or pembrolizumab and/or any of their excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a known history of Human Immunodeficiency Virus (HIV).
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (HCV) (defined as detectable HCV RNA) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
* Liver cirrhosis.
* Has a known history of active TB (Bacillus Tuberculosis).
* Is currently using megestrol acetate or megestrol acetate containing drugs within 10 days of registration.
* Has a history of cerebrovascular accident (CVA), transient ischemic attack (TIA) or carotid artery disease requiring intervention / treatment.
* Has New York Heart Association Class III or IV cardiac disease (Appendix 5) or myocardial infarction within the past 12 months.
* Has known allergy to hyaluronidase.
* Has clinical evidence of Deep Vein Thrombosis (DVT), PE or known thromboembolic event present during the screening period.

  1. Subjects with superficial vein thrombosis are eligible.
  2. Subjects with visceral/splanchnic vein thrombosis are still eligible, if in the opinion of the investigator, the visceral/splanchnic vein thrombosis is primarily associated with the anatomic location of the underlying disease of metastatic pancreatic cancer.
* Active bleeding issues or a pathologic condition that is associated with high risk of bleeding.
* Unable to tolerate low-molecular weight heparin 1 mg/kg as prophylaxis.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-15 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) rate | 2 years
  PFS is calculated as the number of days from date of registration to date of disease progression or symptomatic deterioration, or death due to any cause. PFS will be assessed from date of registration through study closure, up to 24 months.

SECONDARY OUTCOMES:
Overall Survival Rate median | 2 years
  Overall survival is calculated as the number of days from date of registration to date of death due to any cause. Overall survival is assessed from date of registration to study closure, up to 24 months.
Overall Response Rate (ORR) | 2 years
  To determine the overall response rate (ORR) of patients by RECIST v1.1. guidelines, that have at least a 30% reduction in tumor volume on a CT scan. ORR is calculated by adding the complete responses with the partial responses, based on RECIST v1.1, recorded at each disease evaluation for each patient. ORR is assessed from Day 1 of treatment to study closure, up to 24 months.
Number of patients with treatment related adverse events as assessed by CTCAE v5.0 | 2 years
  Adverse events will be assessed using CTCAE v5.0 from Day 1 of study treatment through 30-days past the last study treatment per patient, through study closure, up to 24 months. A measure rate of grade 3 or greater adverse events for patients treated with gemcitabine plus nab-paclitaxel with PVHA and pembrolizumab.

OTHER OUTCOMES:
To evaluate pre-treatment and on-treatment PD-L1 | 2 years
  To measure the ratio of patients with pre-treatment and on-treatment PD-L1 expression.
Evaluate tumor Hyaluronan (HA) levels | 2 years
  Hyaluronan levels will be measured in tumor biopsy samples during each patient's study treatment with data assessed until study closure, up to 24 months. The researcher will count the number of patients that go from Hyaluronan high status to low.
  Evaluate pre-and post-treatment Hyaluronan levels in tumor samples, and correlate with ORR, PFS, and OS.
Change in immune effector cells with treatment | 2 years
  Immunohistochemistry of T-cells and macrophage subsets are measured in tumor tissue samples during each patient's study treatment, with data assessed until study closure, up to 24 months.
  Evaluate pre-and post-treatment immune effector cell levels in tumor samples, and correlate with ORR, PFS, and OS.
Number of patients with additional tissue to cryopreserve | 2 years
  Unused tumor tissue from tumor biopsies obtained during each patients study treatment will be cryopreserved. Evaluate the number of patients with additional tissue available for cryopreservations.
Number of patients with available tumor tissue to create organoid cultures | 2 years
  Unused tumor tissue from tumor biopsies obtained during each patients study treatment will be used to create tumor derived organoids.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Cecchin, MD, Principal Investigator — Yale University